CLINICAL TRIAL: NCT05941091
Title: Effect of the HafifMod Programme for Fluid and Salt Control Guided by Health Belief Model on Interdialytic Weight Gain in Routine Hemodialysis Patients
Brief Title: Effect of the HafifMod Programme on Interdialytic Weight Gain in Hemodialysis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, SALİH GÜLER, Specialist Nurse, Akdeniz University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Sal.h7331
Record Dates: First submitted 2023-06-14; First posted 2023-07-12 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: End-Stage Renal Disease; Hemodialysis; Interdialytic Weight Gain
Keywords: Hemodialysis patients; Fluid control; Salt control; Interdialytic weight
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group or HafifMod Group (Experimental): The HafifMod Programme; It consists of modular education practice and a mobile application offered to HD patients.
  Interventions: Behavioral: HafifMod Programme
- Control group (Active Comparator): Prepared by a dietitian; As a result of the distribution of a printed material called "Nutrition Guide for Dialysis Patients" to the active control group, individuals will be informed about nutrition.
  Interventions: Behavioral: Distribution of printed material

INTERVENTIONS:
Behavioral: HafifMod Programme — MODULAR EDUCATION PROGRAMME: A training program consisting of five modules, shaped by the main headings of fluid and salt control in hemodialysis patients, was created. It is aimed that the patients receive training on a topic each week in a gradual manner. It will be ensured that HD patients can watch the modular training videos prepared in the computer environment on a tablet or computer.
  MOBİLE APPLICATION: Through the mobile application to be developed, the maximum amount of fluid that HD patients should consume per day will be calculated automatically based on their dry weight. In addition, a system will be created where the user can manually enter the amount of fluid consumed daily and add it to the total amount of fluid consumed. In this way, people will be able to learn the amount of fluid they consume daily. In addition, the content of the application will include informative messages in the form of educational short tips and modular training videos.
  Arms: Intervention Group or HafifMod Group
Behavioral: Distribution of printed material — In the study, a general dietary guideline including fluid and salt restriction, which is a printed educational material for the control group, will be used. Thus, it is planned that the participants in the control group will have a guide resource that will enable them to be informed about nutrition. In this way, an educational practice based on the distribution of printed material will be carried out for the control group. Except for the material distribution practice, the routine care procedures the unit will be maintained in the same way, and no different a practice will be made.
  Arms: Control group

SUMMARY:
Haemodialysis (HD) is the most commonly used method among renal replacement therapy options in patients with End Stage Renal Failure. Although one of the most important factors affecting the success of this treatment is compliance with fluid restriction, the rates of non-compliance with fluid control vary between 10-74%. It is understood from the literature that fluid restriction is one of the most difficult areas in compliance with HD treatment. Interdialytic weight gain is the most widely accepted method to assess compliance with fluid control by measuring the amount of fluid accumulated in the body. Thus, studies on this subject have shown that excessive interdialytic weight gain is a common problem in HD patients. It is known that excessive interdialytic weight gain increases the risk of morbidity and mortality in HD patients. The main factors causing interdialytic weight gain are fluid and salt intake between two HD sessions is appears to be. Therefore, it is stated that the easiest solution to control excessive interdialytic weight gain is to reduce fluid and salt intake. However, studies have reported that HD patients have difficulty in adapting to a salt-restricted diet, and in this case, they increase their fluid consumption. Therefore, it is of vital importance that public health nurses carry out interventions to ensure HD patients' compliance with fluid and salt control. In the literature review conducted with this perspective, studies were encountered in which results were obtained that m-health interventions provided a decrease in interdialytic weight gain averages and sodium intake. In this direction, a HafifMod programme based on the use of mobile health technologies was created. The aim of the study is to examine the effect of the LightMod programme for fluid and salt control guided by the Health Belief Model on interdialytic weight gain in routine haemodialysis patients.

DETAILED DESCRIPTION:
Methods such as patient education and self-monitoring have been reported to be effective in ensuring compliance of haemodialysis patients with dietary and fluid restrictions. Methods accepted to be effective in ensuring compliance with fluid restriction include measuring the amount of fluid intake throughout the day, sharing the fluid to be taken during the day, and avoiding salty foods in patients' diets. It is stated that m-Health applications such as recording diet and fluid intake for monitoring and evaluation of nutrition are very useful for self-diet management of dialysis patients. At the same time, it is stated that the training approach based on the delivery of training modules created for the management of chronic diseases through mobile technological tools such as tablet computers has potential benefits.

It is thought that individual beliefs, values and attitudes have a significant impact on the health behaviors of routine HD patients to adapt to fluid and salt restriction.Therefore, interventions within the framework of the HafifMod programme, which will be prepared in line with the Health Belief Model, may be effective in developing positive beliefs, attitudes and behaviours towards fluid and salt control in routine HD patients.

The study is a quasi-randomised active controlled experimental study with single blind (participant) structure. The population of the study consisted of patients receiving routine haemodialysis treatment in the HD unit of Akdeniz University Hospital. According to the days of treatment, there are two separate groups receiving HD treatment 'Monday-Wednesday-Friday' or 'Tuesday-Thursday-Saturday'. As a result of the draw of lots, the groups were divided into two (intervention and active control) according to the days of treatment.Each group is planned to have an equal number of 17 participants. A quasi-randomised controlled study was designed in which sample selection would be made by random sampling method among the intervention and active control groups. This design was based on the principles of the TREND (Transparent Reporting of Evaluation with Nonrandomised Designs) guideline, which is recommended for the design and reporting of quasi-experimental studies.

HafifMod Programme consists of a modular training application and a mobile application offered to HD patients.The implementation period of the HafifMod programme consists of a 3-month period.Repeated measurements will be made for the intervention and active control groups, and a total of four tests will be performed at the 1st, 4th, 8th and 12th weeks.Modular training will be continued for a total of 5 weeks. Patient follow-up will be performed in the remaining weeks. Interdialytic weight gain and monthly serum sodium levels will be monitored at the beginning of each dialysis session. In addition, pre-test and post-test measurements will be performed using the Fluid Control in Haemodialysis Patients Scale and the Beliefs about Dietary Compliance Scale.

ELIGIBILITY:
Inclusion Criteria:

* Those who gained more than 3% of their dry weight in at least one of the interdialytic weight gains covering the four-week period before the start of the study,
* Those who have received routine HD treatment for at least three months,
* Those whose dry weight has been determined,
* Smartphone users,
* Those who do not have severe visual and hearing impairment that would constitute an obstacle to the research,
* Those who are place, time and person oriented,
* Outpatients receiving HD treatment,
* Those with a routine HD program of 3 days and 4 hours a week,
* Those who do not have a psychiatric disorder that would constitute an obstacle to the research.

Exclusion Criteria:

* Those receiving home hemodialysis treatment,
* Those in the home hemodialysis training process,
* Those with plans to make changes to the dialysis center in the next three months from the start of the study,
* Patients who do not undergo ultrafiltration because their urine volume is sufficient.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-10-15 (Estimated); Primary Completion 2024-01-15 (Estimated); Study Completion 2024-10-15 (Estimated)

PRIMARY OUTCOMES:
Interdialytic Weight Gain | 0-3 months (Repeated tests at 1, 4, 8 and 12 weeks)
  H1: Decrease in the mean of interdialytic weight gain- The difference between the weight measured at the entrance to the hemodialysis session and the predetermined dry weight of the patient will be recorded as the interdialytic weight gain value. In addition, a single ramp dialysis scale will be used for weight measurement and the measurements will be recorded in kg. The measurement data obtained during the dialysis sessions within the 3-month research period will be recorded in the 'Session Attendance and Weight Tracking Chart (Chart-1)'.

SECONDARY OUTCOMES:
Fluid Control in Hemodialysis Patients Scale | 0-3 months (Repeated tests at 1 and 12 weeks)
  H1: Increased level of compliance with fluid control- It was developed by Cosar and Pakyuz (2016) to measure the knowledge, behavior and attitudes of hemodialysis patients about fluid restriction. The scale has a total of 24 items and three sub-dimensions.As the score obtained from the scale increases, the compliance of the patients to fluid control also increases. Cronbach alpha internal consistency coefficients of the scale; It is 0.92 for the knowledge sub-dimension, 0.80 for the behavior sub-dimension, and 0.67 for the attitude sub-dimension.
Serum Sodium Level | 0-3 months (Repeated tests at 1, 4, 8 and 12 weeks)
  H1: Decreased serum sodium levels- In order to monitor the blood biochemistry values of all patients who are being treated in the HD unit of Akdeniz University Hospital and to arrange the treatment accordingly, blood samples are taken from the patients on a monthly basis and sent to the Central Laboratory of the Akdeniz University Hospital. In these tests, the serum sodium level is also checked along with other biochemical parameters. Thus, our study will be based on the serum sodium level results obtained from these assays. In our study, the reference range of serum sodium level of Akdeniz University Hospital Central Laboratory, 136-145 mEq/L, will be based on. In addition, serum sodium levels obtained as a result of patient assays will be recorded in the 'Sodium Follow-up Schedule (Schedule-2)'.
Beliefs About Dietary Compliance Scale | 0-3 months (Repeated tests at 1 and 12 weeks)
  H1: Increased levels of perceived benefit for compliance with dietary salt restriction- Beliefs About Dietary Compliance Scale, Bennett et al. (2001) to evaluate the perceptions of benefits and barriers in patients with heart failure in compliance with salt restriction. The Cronbach's alpha coefficients of the developed scale were 0.83 for the benefit sub-dimension and 0.66 for the disability sub-dimension. The first validity and reliability of the Beliefs About Dietary Compliance Scale in Turkey, Oğuz et al. (2010), Cronbach alpha coefficients; Benefit sub-dimension was found to be 0.71, while disability sub-dimension was found to be 0.58.Each sub-dimension in the scale is evaluated separately. A high score from the benefit sub-dimension indicates that the perceived benefit in adhering to a salt-restricted diet is high, while a high score from the barrier sub-dimension indicates that the perceived barriers to adherence to a diet are high.
Beliefs About Dietary Compliance Scale | 0-3 months (Repeated tests at 1 and 12 weeks)
  H1: Decreased levels of perceived barrier to compliance with dietary salt restriction- Beliefs About Dietary Compliance Scale, Bennett et al. (2001) to evaluate the perceptions of benefits and barriers in patients with heart failure in compliance with salt restriction. The Cronbach's alpha coefficients of the developed scale were 0.83 for the benefit sub-dimension and 0.66 for the disability sub-dimension. The first validity and reliability of the Beliefs About Dietary Compliance Scale in Turkey, Oğuz et al. (2010), Cronbach alpha coefficients; Benefit sub-dimension was found to be 0.71, while disability sub-dimension was found to be 0.58. Each sub-dimension in the scale is evaluated separately. A high score from the benefit sub-dimension indicates that the perceived benefit in adhering to a salt-restricted diet is high, while a high score from the barrier sub-dimension indicates that the perceived barriers to adherence to a diet are high.

CONTACTS AND LOCATIONS:
Locations (1):
- Salih Güler, Kepez, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It will not be shared for the purpose of confidentiality and protection of personal data.

REFERENCES:
- [Background] Hong LI, Wang W, Chan EY, Mohamed F, Chen HC. Dietary and fluid restriction perceptions of patients undergoing haemodialysis: an exploratory study. J Clin Nurs. 2017 Nov;26(21-22):3664-3676. doi: 10.1111/jocn.13739. Epub 2017 Mar 22. PMID 28122399